CLINICAL TRIAL: NCT03252405
Title: the Effect of Two Different Method; Mask Ventilation or Intravenous Canulation on Emergence Agitation and Recovery Conditions on Pediatric Adenotonsillectomy
Brief Title: Effect of Induction Method in Post Operative Agitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Kevser Peker, MD, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: emergence agitation
Record Dates: First submitted 2017-08-08; First posted 2017-08-17 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Emergence Agitation
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mask ventilation (Active Comparator): induction is made with mask ventilation
  Interventions: Device: mask ventilation; Device: intravenous cannulation
- intravenous induction (Experimental): induction is made with intravenous cannulation
  Interventions: Device: intravenous cannulation

INTERVENTIONS:
Device: mask ventilation — before intravenous induction, mask application is made. then intravenous cannulation and induction
  Other Names: induction method with mask ventilation
  Arms: mask ventilation
Device: intravenous cannulation — induction is applied by using intravenous cannulation
  Other Names: induction method with intravenous cannulation

SUMMARY:
To compare the effect of two different induction method; mask ventilation and intravenous cannulation on emergence agitation on pediatric adenotonsillectomy

DETAILED DESCRIPTION:
Many things cause emergence agitation after operations on pediatric population. This research aims determine which method, mask ventilation or intravenous cannulatin is more effective on emergence agitation

ELIGIBILITY:
Inclusion Criteria:

* pediatric adenotonsillectomy

Exclusion Criteria:

* patients with neurological, hepatic, renal disorders and using any drugs

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
assess changing in pediatric agitation/ emergence delirium scale(PAED) scores | postoperative first hour
  to asses change of intensity of postoperative emergence agitation/ delirium (PAED) by using pediatric agitation emergence delirium scale with scores. to assess changing PAED scores at one hour after transfer into the post anesthesia care unit.

SECONDARY OUTCOMES:
FLACC (face, legs,activity, cry, consolobility) | postoperative first hour
  to asses postoperative pain intensity with scores by FLACC (face, legs,activity, cry, consolobility) scale after transfer into the post anesthesia care unit

CONTACTS AND LOCATIONS:
Overall Officials: kevser peker, Principal Investigator — Ahi Evran University Education and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Dışkapı Yıldırım Beyazıt Education and research hospital, Ankara
  - Ahi evran university education and research hospital, Kırşehir

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peker K, Polat R. Effects of intravenous and mask induction on post-operative emergence delirium in pediatric patients undergoing tonsillectomy with or without adenoidectomy. Ir J Med Sci. 2020 Aug;189(3):1061-1068. doi: 10.1007/s11845-020-02197-4. Epub 2020 Feb 11. PMID 32048203